CLINICAL TRIAL: NCT02456129
Title: An Open-label Study to Evaluate the Effect of Repeated Oral Administration of 200 mg Itraconazole(ITZ) Given Once Daily Over 14 Days on the Single Oral Dose Pharmacokinetics of Vilaprisan (BAY1002670) as Well as Assessment of Absolute Bioavailability Using a Single Intravenous Microtracer Dose of [14C]Vilaprisan in Healthy Postmenopausal Women
Brief Title: Study in Postmenopausal Women to Investigate the Drug-drug Interaction (DDI) Between Itraconazole(ITZ) and Orally Administered Vilaprisan; Absolute Bioavailability Using Intravenous Microtracer Dose of [14C]Vilaprisan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 15250; 2014-004929-41 (EudraCT Number)
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Clinical Trial, Phase I
Keywords: Clinical Trial, Phase I
MeSH Terms: interventions — vilaprisan; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vilaprisan + Itraconazole (Experimental): Vilaprisan (BAY1002670)
  Interventions: Drug: Vilaprisan (BAY1002670); Drug: [14C] Vilaprisan; Other: Itraconazole(ITZ)

INTERVENTIONS:
Drug: Vilaprisan (BAY1002670) — single oral doses of 4 mg tablet Vilaprisan, administered once without the comedication of ITZ (period 1) and once with the comedication of ITZ (period 2)
Drug: [14C] Vilaprisan — an intravenous microtracer dose of [14C]Vilaprisan administered together with the 1st single oral dose of Vilaprisan
Other: Itraconazole(ITZ) — Itraconazole(ITZ) 200 mg as solution, once daily for 14 days

SUMMARY:
This is a study in postmenopausal women to investigate the Drug-drug interaction (DDI) between itraconazole(ITZ) and orally administered vilaprisan; absolute bioavailability using intravenous microtracer dose of [14C]vilaprisan.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI): 18 ≤ BMI ≤ 32 kg/m²
* Postmenopausal state revealed by:

Medical history, if applicable (natural menopause at least 12 months prior to first study drug administration; or surgical menopause by bilateral ovariectomy at least 3 months prior to first study drug administration), in addition: in women < 65 years old, follicle stimulating hormone (FSH) > 40 IU/L

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination or effects of the study drugs will not be normal
* Known or suspected liver diseases
* Clinically relevant findings(e.g. blood pressure, electrocardiogram(ECG); physical and gynecological examination, laboratory examination)

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve [AUC(0-11d)] after single oral dose of vilaprisan with and without ITZ. | up to 14 days
Maximum plasma concentration (Cmax) after single oral dose of vilaprisan with and without ITZ. | up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] Schultze-Mosgau MH, Hochel J, Prien O, Zimmermann T, Brooks A, Bush J, Rottmann A. Characterization of the Pharmacokinetics of Vilaprisan: Bioavailability, Excretion, Biotransformation, and Drug-Drug Interaction Potential. Clin Pharmacokinet. 2018 Aug;57(8):1001-1015. doi: 10.1007/s40262-017-0607-4. PMID 29330782